CLINICAL TRIAL: NCT04579796
Title: The Accuracy of Ultrasound in the Detection of Placenta Site in the First Trimester When Compared to Hysteroscopy in Early Abortions
Brief Title: The Accuracy of Ultrasound in the Detection of Placenta Site in the First Trimester.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Doctor, Assaf-Harofeh Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: # 0178-19
Record Dates: First submitted 2020-08-26; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Placenta; Implantation

STUDY DESIGN:
Masking Description: The performer of the hysteroscopy will not be aware of the result of the ultrasound exam
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women with first trimester missed abortion (Experimental)
  Interventions: Other: ultrasound exam; Procedure: hysteroscopy diagnostic

INTERVENTIONS:
Other: ultrasound exam — An abdominal ultrasound exam to assess the placenta implantation site.
Procedure: hysteroscopy diagnostic — Diagnostic hysteroscopy to asses the placenta implantation site.

SUMMARY:
The investigators speculate that ultrasound examination in the first trimester can accurately detect placental location. By performing both transabdominal ultrasound and later hysteroscopy on women with a first trimester missed abortions and comparing the ultrasound findings to those of the hysteroscopy the investigators will evaluate the performance of the ultrasound in detecting the placenta location.

DETAILED DESCRIPTION:
All women with a first trimester missed abortion who will sign an informed consent form will undergo an ultrasound examination. During the examination, the operator will assess the location of the placenta/sac insertion. After the performance of the ultrasound, the women will undergo hysteroscopy with a different operator who will be blinded to the results of the previous exam result. During the hysteroscopy the second operator will assess again the location of the sac insertion .The investigatorswill then compare the results of the two tests using the histeroscopy as the gold standard and evaluate the performance of abdominal ultrasound exam in the evaluation of placenta/ sac inserion.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women .
* Clinical diagnosis of first trimester spontaneous abortion.

Exclusion Criteria:

* viable pregnancy
* women below 18 years
* women with chronic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of placental site/ gestational sac implantation with ultrasound in the first trimester | up to 12 weeks
  Transabdominal ultrasonography detection of gestational sac insertion location will be compared with gestational sac location diagnosed with hysteroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Asaf ha Rofeh, MC, Zrifin, Israel